CLINICAL TRIAL: NCT03054701
Title: The Acute Effects of Hip and Knee Exercises on Pain Sensitivity in Young Adult Females With Long-standing Patellofemoral Pain - a Randomized Crossover Study.
Brief Title: Effects of Hip and Knee Exercises on Knee Pain in Young Adult Females With Long-standing Patellofemoral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Michael Skovdal Rathleff, Associate Professor, Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: N-20160058
Record Dates: First submitted 2017-02-09; First posted 2017-02-16 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral pain; PFP; PFPS
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: After providing informed consent the participants will determine which is their most painful knee. This limb will be marked and it will serve as the test limb throughout the study protocol. At the first step of the protocol the participants will be baseline tested with handheld and cuff pressure algometer. Secondly, participants will be randomized to either a hip or a knee exercise. Thirdly, participants will undergo the testing-procedure for the second time. Fourthly, participants will perform exercise focusing on the other joint (hip or knee). Finally, participants will undergo the testing-procedure for the last time. In order to avoid any carryover effect from the testing procedure, there will be at least 15-minutes between each of the three test sessions.
Who Masked: Participant, Outcomes Assessor
Masking Description: The outcome assessor will be blinded to the order of the exercises and the participants will be blinded to the study-hypothesis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sidelying hip abduction exercise (Experimental): Participants will be lying on the side with both legs stretched and with their head resting on a pillow. Participants will be allowed to place their hand in front of them to fixate their body and maintain balance. The participants will be instructed to abduct their hip to 45 degrees and return to the resting position afterwards. An elastic band will be used as resistance. This exercise will be applied only on the test limb. A digital metronome will be used to maintain the pace during the exercise.
  Load: 12 repetition maximum; Nr. of repetition: 12; Nr. of sets: 3; Rest between sets: 120 seconds; Time under tension: 8 seconds; Distribution of load: Concentric (3 seconds), Eccentric (3 seconds), Isometric (2 seconds).
  Interventions: Other: Hip specific resistance exercise
- Sitting knee extension exercise (Active Comparator): Participants will be seated at the end of an examination couch with the hip and knee relaxed in a 90 degrees angel. Participants will be allowed to place their hands on the side of the couch and the stabilizing foot may have contact with the floor. The participants will be instructed to extend their knee to a 180-degree angle and return to the resting position afterwards. An elastic band will be used as resistance. This exercise will be applied only on the test limb. A digital metronome will be used to maintain the pace during the exercise.
  Load: 12 repetition maximum; Nr. of repetition: 12; Nr. of sets: 3; Rest between sets: 120 seconds; Time under tension: 8 seconds; Distribution of load: Concentric (3 seconds), Eccentric (3 seconds), Isometric (2 seconds).
  Interventions: Other: Knee specific resistance exercise

INTERVENTIONS:
Other: Hip specific resistance exercise — Hip specific resistance exercise
  Arms: Sidelying hip abduction exercise
Other: Knee specific resistance exercise — Knee specific resistance exercise
  Arms: Sitting knee extension exercise

SUMMARY:
Patellofemoral pain (PFP) is highly prevalent in both adolescent and adult populations and as much as 91% of those affected experience ongoing knee pain for up to 20 years after the initial diagnosis.

Exercise-based treatment focusing on strengthening the muscles around the hip and knee is usually effective when treating patient with PFP. However, this approach has proven ineffective in a subgroup of females who have suffered from PFP for multiple years.

This group was found to have a significantly lower tolerance for pressure stimuli compared to healthy controls. This indicating that central mechanisms within the nervous system rather than the problem being the knee itself.

Exercising a non-painful muscle distant to a painful part of the body has previously been effective in deceasing pain in affected area. This mechanism has been investigated in patients with long-standing musculoskeletal pain as well as healthy populations.

Related research has suggested that a possible link between patients perception of painful stimuli an the pain-reducing effect of exercise exists. As such, patients witch experienced a pain reducing effect of exercise was found to be able to tolerate more pain than before the intervention.

The aim of this study is to assess if exercising a distant non-painful muscle around the hip has a larger acute pain-reducing effect on knee pain compared to knee specific exercises in female patients with long-standing PFP.

DETAILED DESCRIPTION:
Background: Patellofemoral pain (PFP) has a high prevalence in both adolescent and adult populations (7% and 15%) and as much as 91% of those affected experience ongoing knee pain for up to 20 years after the initial diagnosis. Exercise-based treatment focusing on strengthening the muscles around the hip and knee is usually effective when treating patient with PFP. However, this approach has proven ineffective in a subgroup of females with long-standing PFP. This group was found to have altered condition pain modulation indicating facilitated central mechanisms. A localized analgesic effect by exercising a distant non-painful muscle has been observed previously in patients with long-standing musculoskeletal pain. This is known as exercise induced hypoalgesia. In relation, an increased condition pain modulation was found to be a predictor for an increase in the effect of exercise induced hypoalgesia, indicating a link between the two mechanisms. The aim of this study is to assess if exercising a distant non-painful muscle around the hip has a larger acute analgesic effect on localized knee pain compared to knee specific exercises in female patients with long-standing PFP.

Study design: This study is a randomized, controlled, participant and assessor blinded crossover study. The study will be conducted at the Research Unit of General Practice in Aalborg. Reporting of the study will follow the CONSORT guidelines for randomized trials of Non-pharmacologic Treatment.

Method: Thirty women between the age of 20 and 25 with current knee pain which they have experienced ongoing or recurrent for a duration of 5 years will be randomized to either a knee or hip specific resistance exercise as their first intervention. After a washout period of 15 minutes, the participant will perform the other exercise. The participants will undergo a test-procedure before the first exercise, between the exercises and after the final exercise. The test-procedure consist of handheld pressure algometry and cuff pressure algometry assessing pain pressure threshold, pain detection threshold and pain tolerance threshold. Condition pain modulation and temporal summation of pain will be assessed by cuff algometry. In order to assess knee pain in relation to the exercises, the participants will be asked to rate their knee pain before and after each exercise set. The primary outcome will be pain pressure threshold assessed by handheld pressure algometry at the center of patella of the test limb.

Recruitment: A random sample of participants from the APA2011 cohort who experience ongoing PFP in 2016 will be invited to participate in this study. The participants will be contacted by telephone and invited to participate in the study. Verbal information regarding the study will be provided over the phone and written material will be send by e-mail. In case the cohort provide an insufficient number of participants, patients from general practice will be sought out and invited to participate. This process will be done in collaboration with general practice clinics in the area. If the combination of the above-mentioned strategies does not provides the required number of participants, online social-medias like Facebook and Twitter will be used as a mean to obtain a sufficient number of participants.

Allocation sequence: The participants will be randomized to do either sitting knee extension or sidelying hip abduction first. A computer generated allocation sequence will be conducted at www.random.org by an independent researcher. This individual will put slips of paper, which says either "Hip" or "Knee" into opaque sealed envelopes. The envelopes will be marked with sequential numbers. When the first participant have underwent the baseline testing he or she will be assigned the ID number 1 (ID1). After completing the baseline test this participant will proceed to the exercise room where the exercise instructor will be waiting. The exercise instructor will then select the envelope marked "ID1" and note if the participant was assigned to the hip or knee exercise as the first exercise.

Familiarization session: Before each exercise, the load at which the participants can do exactly 12 repetitions will be established by using elastic band with different elastic abilities. This will also work as a familiarization session where the participants can get to know the exercises. For the familiarization session, a black elastic band will be used as default for the sitting knee extension exercise, whereas a yellow elastic band will be used in the sidelying hip abduction exercise. If the participants are capable of performing more or less than 10-12 repetitions with the default elastic band, the length or color will be changed to ensure the participants exercise at 12RM.

Precautions: Participants will be asked to withstand from caffeine, alcohol, nicotine and physically exhausting activities for up to 24 hours before undertaking the study protocol as these have been shown to have a dampening effect on pain. Due to the nature of the study, participants are encouraged to withstand from taking any analgesics on the day for undergoing the study protocol.

Data analysis: A preliminary analysis to see if order of exercise has an effect on the results will be conducted. To investigate if there is any statistically significant difference in PPT, pain detection threshold (PDT) and pain tolerance threshold (PTT) and VAS scores measured at the three time-points, a repeated measure analysis of variance (ANOVA) will be undertaken if data is found to be normally distributed. If data is not normally distributed the Kruskal-Wallis test will applied instead. This data will be presented with a mean, a standard deviation, an f-value and a p-value. For the PPT, PDT and PTT a mean difference of 50 kPa is considered to be clinically relevant.

In addition, the association between knee pain intensity at baseline testing and EIH response for hip versus knee exercises will be investigated. By doing this test it will be possible to assess if those with greater knee pain intensity has a larger EIH response from hip exercises compared to knee exercises.

To assess flare up in pain during exercise the mean change in numeric pain ratings from start to finish of each set within each exercise (hip or knee) will be calculated.

To investigate if there is any correlation between handled PPT measured at the three sites (center of patella on the test limb, the belly of the m. tibialis anterior muscle og the test limb and the epicondyle of the contralateral elbow) a test for correlation will be conducted.

In order to examine if the flare up in pain during exercise behave the same way as TSP, a test for correlation between these two variables will conducted.

Sample size: A group of 10 healthy subjects volunteered to participate in a pilot study prior to recruitment of the current study. Data regarding handheld PPT measured at the center of patella was used to calculate the sample size required to power the study. The mean difference between handheld PPT after hip exercise and after knee exercise within the group was 44 kPa with a corresponding standard deviation of 80 kPa. These data was used in a two-sided power analysis for two paired means which was conducted in STATA. With a significant level of 0.05 and the power set to 0.8, a minimum of 28 participants would be required to power the study. However, 30 participants will be included in order to insure the study is adequately power in case of missing data due to system malfunction or if the effects size turns out to be lower than the anticipated 0.55.

This randomized study is embedded within a larger cross-sectional study which is approved by the ethical committee under the same approval number (N-20160058). This can be accessed on clinicaltrials.gov under the title "Pain mechanisms in Young Adolescent Females With Longstanding Patellofemoral Pain" with Dr. Sinead Holden as the primary investigator.

ELIGIBILITY:
Inclusion Criteria:

* Participants with PFP are required to have current non-traumatic anterior or retropatellar knee pain which they have experienced ongoing or recurrently for a duration of at least 5 years.
* At least two of the following daily activities should provoke knee-related symptoms: prolonged sitting or kneeling, squatting, running, hopping, or stair walking, tenderness on palpation of the patella or double leg squatting.
* Worst pain during the previous week have to be of more than 3 cm on a 10-cm visual analog scale (VAS).

Exclusion Criteria:

* Patients who have sustained a traumatic injury to the hip, knee, ankle or the lumbar spine within the past 3 month will be excluded.
* Other identifiable knee conditions in isolation (that is, not occuring concurrently with PFP. As an example, if the subject has isolated patellar tendinopathy they will be excluded. If the subject has PFP and concurrent pain at the patellar tendon, they will be included).
* Individuals with rheumatoid arthritis, knee joint effusion, self-reported patellofemoral instability, known malign conditions, neurological disease or previously knee surgery will be excluded as well.
* In cases with suspicion of serious pathology a rheumatologist will be consulted.

Ages: 20 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain pressure threshold (PPT) at the center of patella. | This will be assessed at 1) baseline, 2) approximately 5 minutes after the first exercise intervention (hip or knee) and 3) approximately 5 minutes after the second exercise intervention (hip or knee).
  The acute effect of hip versus knee exercises on PPT at the center of patella will be compared. These measures will be taken from the test limb. PPT is defined as the point where pressure becomes painful and will be assessed by handheld pressure algometry (SOMEDIC Electronics, Solna, Sweden). The pressure will be applied with at a rate of 30 kPa/s at a perpendicular angle, to a 1cm2 area on the skin surface. Subjects will be given a handheld switch and will be instructed to press it as soon as the stimulus changes from pressure to pain. PPT will be measured twice at each time-point and the average will be calculated and used for the analyses. A mark will be drawn on the center of patella to make sure the two measures are taken from the same site. There will be a 30-second break between each measurements.

SECONDARY OUTCOMES:
Change in PPT at the muscle belly of the m. tibialis anterior. | This will be assessed at 1) baseline, 2) within 20 minutes after completing the first exercise intervention (hip or knee) and 3) within 20 minutes after completing the second exercise intervention (hip or knee).
  The acute effect of hip versus knee exercises on PPT at the muscle belly of the m. tibialis anterior will be compared. These measures will be taken from the test limb. PPT is defined as the point where pressure becomes painful and will be assessed by handheld pressure algometry (SOMEDIC Electronics, Solna, Sweden). The pressure will be applied with at a rate of 30 kPa/s at a perpendicular angle, to a 1cm2 area on the skin surface. Subjects will be given a handheld switch and will be instructed to press it as soon as the stimulus changes from pressure to pain. PPT will be measured twice at each time-point and the average will be calculated and used for the analyses. A mark will be drawn on the muscle belly of the m. tibialis anterior to make sure the two measures are taken from the same site. There will be a 30-second break between each measurements.
Change in PPT at the lateral epicondyle on the contralateral elbow. | This will be assessed at 1) baseline, 2) within 20 minutes after completing the first exercise intervention (hip or knee) and 3) within 20 minutes after completing the second exercise intervention (hip or knee).
  The acute effect of hip versus knee exercises on PPT at the lateral epicondyle on the contralateral elbow will be compared. These measures will be taken from the contralateral elbow of the test limb. PPT is defined as the point where pressure becomes painful and will be assessed by handheld pressure algometry (SOMEDIC Electronics, Solna, Sweden). The pressure will be applied with at a rate of 30 kPa/s at a perpendicular angle, to a 1cm2 area on the skin surface. Subjects will be given a handheld switch and will be instructed to press it as soon as the stimulus changes from pressure to pain. PPT will be measured twice at each time-point and the average will be calculated and used for the analyses. A mark will be drawn on the lateral epicondyle on the contralateral elbow to make sure the two measures are taken from the same site. There will be a 30-second break between each measurements.
Change in pain detection threshold (PDT) measured with cuff pressure allometry at the lower leg of both limbs. | This will be assessed at 1) baseline, 2) within 20 minutes after completing the first exercise intervention (hip or knee) and 3) within 20 minutes after completing the second exercise intervention (hip or knee).
  The cuff will inflate with 1 kPa per second and the participants are instructed to start rating their pain on the electronic VAS as soon as the sensation of pressure becomes painful (pain detection threshold).
Change in pain tolerance threshold (PTT) measured with cuff pressure allometry at the lower leg of both limbs. | This will be assessed at 1) baseline, 2) within 20 minutes after completing the first exercise intervention (hip or knee) and 3) within 20 minutes after completing the second exercise intervention (hip or knee).
  The cuff will inflate with 1 kPa per second and the participants are instructed to start rating their pain on the electronic VAS as soon as the sensation of pressure becomes painful. Participants are instructed to press the release button when the pain becomes intolerable (pain tolerance threshold).
Change in temporal summation of pain assessed by cuff pressure allometry at the lower leg of the test limb. | This will be assessed at 1) baseline, 2) within 20 minutes after completing the first exercise intervention (hip or knee) and 3) within 20 minutes after completing the second exercise intervention (hip or knee).
  The cuff will apply 10 repetitive stimulus at 100% of the PTT measured by the cuff algometer on the test limb. Each stimulus has a duration of 1 second followed by 1 second where the cuff is deflated. The participant will be asked to rate the pain intensity on an electronic VAS continuously throughout the test. The cuff-system software will automatically identify the highest recorded VAS within each of the 1 second deflations.
Change in condition pain modulation assessed by cuff pressure allometry at the lower leg of the test limb. | This will be assessed at 1) baseline, 2) within 20 minutes after completing the first exercise intervention (hip or knee) and 3) within 20 minutes after completing the second exercise intervention (hip or knee).
  Data on PDT and PTT from the contralateral limb will be used to calibrate the cuff system before this test. The cuff on the contralateral limb will inflated to 70% of the PTT measured from the contralateral limb. Participants are instructed to ignore this pressure an to only focus on the test limb. As before, the cuff on the test limb will inflate with 1 kPa per second and the participants are instructed to start rating their pain on the electronic VAS scale as soon as the sensation of pressure becomes painful (PDT). Participants are instructed to press the release button when the pain becomes intolerable (PTT).
Change in self-reported pain before and after each exercise set reported on a numeric pain rating scale (NPRS). | This will be assessed during the first exercise intevention (hip or knee) and approximately 30 minutes after, during the second exercise intervention (hip or knee).
  Participants will be asked to rate their knee pain intensity right before and immediately after each of the three sets within each exercise. The mean difference between the before and after assessments will be calculated and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Rathleff, PhD, Study Director — Aalborg University
Locations (1):
- Research Unit For General Practice in Aalborg, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No
IPD data will be available on request after manuscript has been published.